CLINICAL TRIAL: NCT04430543
Title: Addressing Problem Drinking From the Bottom-Up: An Investigation of the Neural and Behavioral Effects of Cognitive Bias Modification (CBM)
Brief Title: Neural and Behavioral Effects of Cognitive Bias Modification (CBM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Kelli Tahaney, Principal Investigator, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4633E; 1F31AA025522-01A1 (NIH)
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Alcohol Drinking
Keywords: motivation; alcohol-related disorders; self-control
MeSH Terms: conditions — Alcohol Drinking; Alcohol-Related Disorders; Self-Control

STUDY DESIGN:
Intervention Model Description: There will be 2 groups- treatment group and control group. Both groups will receive a web-based motivational intervention then will be randomized to Cognitive Bias Modification or Sham (control) training. Participants will complete a total of 5 sessions of CBM or Sham over the course of a week.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBM Group (Experimental): This group will receive Cognitive Bias Modification training
  Interventions: Behavioral: Cognitive Bias Modification
- Control Group (Sham Comparator): This group will receive Sham (control) training
  Interventions: Behavioral: Sham Training

INTERVENTIONS:
Behavioral: Cognitive Bias Modification — CBM sessions are computer tasks that take 15 minutes each. CBM is similar to an alcohol approach avoidance task (AAT) in that they will involve moving their mouse forward to simulate an avoidance/push response and backward to simulate an approach/pull response in response to alcohol and neutral stimuli depending on photograph orientation. Photos will get larger as if coming toward the participant when "pulled" and will get smaller as if moving away when "pushed". CBM will involve pushing 90% of alcohol stimuli (pulling 10%) and pulling 90% of neutral stimuli (pushing 10%).
  Arms: CBM Group
Behavioral: Sham Training — Sham training sessions are computer tasks that take 15 minutes each. Sham training is similar to an alcohol approach avoidance task (AAT) in that they will involve moving their mouse forward to simulate an avoidance/push response and backward to simulate an approach/pull response in response to alcohol and neutral stimuli depending on photograph orientation. Photos will get larger as if coming toward the participant when "pulled" and will get smaller as if moving away when "pushed". Sham training will involve pushing and pulling 50% of each type of stimuli (alcohol and neutral)
  Arms: Control Group

SUMMARY:
This study seeks to better understand mechanisms of behavior change for heavy drinkers who are interested in changing their drinking. The study will examine the effects of CBM as an adjunctive treatment on neurocognitive processes related to alcohol use in a sample of heavy/at-risk drinkers using functional magnetic resonance imaging (fMRI). The primary aim of this project is to examine the effects of CBM on neurocognitive approach tendencies and control processes, among heavy/at-risk drinkers interested in changing their alcohol use. As a secondary aim, this project will investigate associations between neural and cognitive changes and changes in alcohol use to better understand how CBM might lead to successful changes in drinking behavior. Either CBM (treatment group) or sham computer task (control group) will be paired with a motivational web-based intervention for alcohol use. Brain activity will be measures twice via fMRI--pre-treatment and 1-week post-treatment. The experimental tasks completed in the fMRI scans include 2 alcohol cue reactivity (CR) tasks--one standard and one in which participants are told to either inhibit (INHIBIT) or engage in (INDULGE) their reaction to images of alcohol and neutral beverages. Follow-up drinking behavior will be measured also at 1-week and online via 1- and 6-month follow-ups. Brain activity at baseline and follow-up will be measured in pre-defined regions of interest including amygdala, NAcc, mPFC, and dlPFC. It is hypothesized that the CBM group will exhibit changes in approach biases as exhibited by reductions in brain activity in the amygdala, NAcc, mPFC in response to alcohol cues in both CR tasks (alcohol CR, INDULGE CR, and INHIBIT CR) compared to sham. In addition, those in the CBM group will show increased dlPFC brain activity during alcohol CR and INHIBIT trials of the cued-CR task as evidence strengthened control abilities in response to alcohol cues. Finally, as a secondary hypothesis, those in the CBM group will show greater reductions in drinking and craving at follow-up.

DETAILED DESCRIPTION:
Forty heavy/at-risk drinkers (ages 18-34) who report an interest in changing their drinking behavior will be recruited for this proposed project. "Interest" will be operationalized as an affirmative answer on an item adapted (for past-month) from the CAGE questionnaire: "In the past month, have you felt you should cut down or stop drinking?" (Mayfield, McLeod, & Hall, 1974). Heavy/at-risk drinking will be defined in terms of consumption (7+/14+ drinks per week and/or 3+/4+ drinks on one occasion over the past week for women and men, respectively; USDHHS, 2005) and score on the Alcohol Use Disorders Identification Test (AUDIT score of 8-19; Babor, Higgins-Biddle, Saunders, & Monteiro, 2001). A score between 8-19 on the AUDIT is indicative of heavy use while scores 20 and above are indicative of a more severe alcohol use disorder (i.e., "dependence", DSM-IV; APA, 2013; APA, 2000). Participants will be recruited through online advertisements on Craigslist, social media websites, and "Quickie Job Board" listings on student websites as well as via flyers in community and student health centers. Upon responding to advertisements participants will be administered a phone screen or complete online screening survey to determine study eligibility.

If eligible, baseline assessments will be administered at an in person appointment, including self-report assessments about alcohol use, drug use, consequences, and alcohol craving. Participants will complete a baseline fMRI scan, which involves administration of two versions of an alcohol cue reactivity (CR) task. Both CR tasks administered in the scanner will consist of a block design. The first alcohol CR task consists of two types of blocks-1) alcohol and 2) neutral beverage (i.e., soft drinks, juice, water). Subjects will be presented with 40 alcohol images and 40 neutral beverage images, respectively. The second task, the cued-CR task, involves 3 blocks utilizing the same images as the alcohol-CR task. Subjects will receive instructions regarding their reaction to the photos-1) INHIBIT CR (alcohol images), 2) INHIBIT NEUTRAL (neutral beverage images), and 3) INDULGE CR (alcohol images). More specifically, participants will be given the instruction to imagine each image is available to them and to either inhibit their natural reaction to the images presented (alcohol in one block, neutral beverages in another block) or think about the possibility of consuming, in this moment, each (alcohol-containing) beverage shown. This task was inspired by fMRI studies using CR tasks and cognitive restraint strategies to inhibit cravings for food and/or alcohol (Naqvi et al., 2015; Yokum & Stice, 2013). For both tasks, each image will be presented for 4 seconds followed by a 2 second inter-image interval. Participants will be asked to rate their level of craving after each block for the first task only. Following this baseline scan, participants will complete a brief web-based intervention for alcohol use, Rethinking Drinking: Alcohol and Your Health (NIAAA, 2015), and will subsequently be randomized to either cognitive bias modification (CBM) or sham training. They will complete the first session of either CBM or sham training after randomization as well as an additional 4 CBM/sham sessions at home (via web) over one week following baseline. Participants will return to the lab one-week following their baseline appointment. At follow-up assessment, participants will complete all baseline assessment measures in addition to a second fMRI session consisting of the same CR tasks. Finally, participants will be emailed a link to a web-based survey at 1- and 6-months following baseline to assess drinking behavior. Data analysis will employ region of interest (ROI) analysis. Predefined ROIs include the bilateral amygdala, nucleus accumbens (NAcc), and dorsolateral and medial prefrontal cortex (dlPFC and mPFC). Anatomical ROIs will be generated using the Wake Forest University (WFU) Pickatlas automatic anatomical labeling tool (Maldjian, Laurienti, Kraft, & Burdette, 2003) available for SPM. The analytic plan for testing study hypotheses are as follows: Primary Aim 1-For the alcohol CR task, two within subject contrasts will be calculated-1] alcohol CR > neutral CR pre-CBM/sham and 2] (alcohol CR > neutral CR) pre-CBM/sham - (alcohol CR > neutral CR) post-CBM/sham-in pre-defined ROIs. Primary Aim 2-as with the alcohol CR task, the within subject contrasts will be 1] INDULGE CR > INHIBIT CR pre-CBM/sham and 2] (INDULGE CR > INHIBIT CR) pre-CBM/sham - (INDULGE CR > INHIBIT CR) post-CBM/sham. Similar within subject contrasts will be explored for INHIBIT CR and INHIBIT NEUTRAL CR as a control. T-tests will be used to compare within subject contrasts for each task as well as to compare between-group contrasts (i.e., alcohol CR and INHIBIT CR pre-and post- CBM/sham). Secondary Aim: Correlations will be run to determine whether BL BOLD activity in each ROI significantly correlate with behavioral measures for both BL and 1-week follow-up. For significant correlations, pre- and post-CBM/sham difference scores will be calculated for behavioral measures and then correlated with significant BOLD contrasts representing change in neural activity.

ELIGIBILITY:
Inclusion Criteria:

* current hazardous drinking (score of 8+ on USAUDIT-C)
* interest in changing drinking
* English-speaking
* able to provide informed consent

Exclusion Criteria:

* Score of 25+ on USAUDIT
* current or past treatment for alcohol or drug use
* lifetime diagnosis of other substance use disorder
* self-reported weekly or more other drug use as indicated on the NIDA-modified Alcohol, Smoking, and Substance Involvement Screening Test
* history of head injury or loss of consciousness
* lifetime diagnosis of bipolar disorder, psychotic symptomatology, organic mental disorder, seizure disorder, or central nervous system disease
* pregnancy
* current use of psychotropic medication
* history of delirium tremens and/or seizures as a result of alcohol withdrawal
* contraindications to fMRI (claustrophobia, pregnancy, metal, pacemaker, etc.).

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
BOLD signal change in ROIs (amygdala, NAcc, mPFC, dlPFC) during alcohol cue-reactivity | 1-week
  decreased signal indicates better outcomes for amygdala, NAcc, and mPFC; increased signal indicates better outcomes for dlPFC
BOLD signal change in ROIs (amygdala, NAcc, mPFC, dlPFC) during INHIBIT cue-reactivity | 1-week
  decreased signal indicates better outcomes for amygdala, NAcc, and mPFC; increased signal indicates better outcomes for dlPFC
BOLD signal change in ROIs (amygdala, NAcc, mPFC) during INDULGE cue-reactivity | 1-week
  decreased signal indicates better outcomes for amygdala, NAcc, and mPFC

SECONDARY OUTCOMES:
Drinking Behavior | 1-week
  Daily Drinking Questionnaire quantity item "most drinks on one occasion"; range 0-31; higher score = more drinking/worse outcome
Drinking Behavior | 1-month
  Daily Drinking Questionnaire quantity item "most drinks on one occasion"; range 0-31; higher score = more drinking/worse outcome
Drinking Behavior | 6-months
  Daily Drinking Questionnaire quantity item "most drinks on one occasion"; range 0-31; higher score = more drinking/worse outcome
Alcohol Craving | 1-week
  Score on Desire for Alcohol Questionnaire; range = 14-98; higher scores reflect higher desire for alcohol (worse outcome)
Alcohol Craving | 1-month
  Score on Desire for Alcohol Questionnaire; range = 14-98; higher scores reflect higher desire for alcohol (worse outcome)
Alcohol Craving | 6-months
  Score on Desire for Alcohol Questionnaire; range = 14-98; higher scores reflect higher desire for alcohol (worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Rajen Kilachand Center for Integrated Life Sciences and Engineering at Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No